CLINICAL TRIAL: NCT06922227
Title: Perioperative Hemodynamic and Respiratory Changes During Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Combined With Cytoreductive Surgery
Brief Title: HIPEC Surgery and Hemodynamics
Status: Not yet recruiting | Type: Observational
Sponsor: Miray Gözde Özdemir (Other Government)
Responsible Party: Sponsor-Investigator, Miray Gözde Özdemir, Anesthesiology and Reanimation specialist / Doctor, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Other Study IDs: 530
Record Dates: First submitted 2025-03-20; First posted 2025-04-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Hemodynamics; Cytoreductive Surgery; Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Keywords: HİPEC; cytoreductive surgery; Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients who will undergo HIPEC with cytoreductive surgery

SUMMARY:
Hyperthermic Intraperitoneal Chemotherapy (HIPEC) involves the intraoperative administration of heated chemotherapeutic agents into the abdominal cavity following cytoreductive surgery (CRS). The increasing use of CRS combined with HIPEC has introduced certain procedural and physiological considerations that distinguish it from other surgical interventions, posing unique challenges for researchers and clinicians alike.

Despite advancements in surgical and anesthetic techniques, this combined approach is frequently associated with significant hemodynamic instability, coagulation abnormalities, respiratory complications, and nutritional imbalances.

The study aims to contribute to the existing body of knowledge by examining the physiological alterations induced by HIPEC, thereby offering practical insights and guidance for investigators involved in the management and study of this complex therapeutic modality.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old Patients planned to undergo cytoreductive surgery with hyperthermic intraperitoneal chemotherapy
* ASA II-III-IV physical class

Exclusion Criteria:

* <18 years
* Emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who are scheduled for cytoreductive surgery with hyperthermic intraperitoneal chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
physiological parameter ; heart rate | Intraoperatively
  HIPEC is usually the application of chemotherapy that lasts between 45 and 90 minutes after the end of cytoreductive surgery. During HIPEC application (45-90 minutes), Heart rate: will be recorded every 10 minutes as beats / minute.
physiological parameter; systolic/diastolic blood pressure | Intraoperatively
  Systolic/diastolic blood pressure will be recorded in mmHg every 10 minutes.
physiological parameter; SpO2 | Intraoperatively
  SpO2 will be recorded as percent every 10 minutes.
anesthesia device measurement parameter; EtCo2 | Intraoperatively
  EtCo2 will be recorded every 10 minutes as mmHg.
anesthesia device measurement parameter; Pmax | Intraoperatively
  Pmax will be recorded as cmH2O every 10 minutes.

SECONDARY OUTCOMES:
Preoperative data | 24 hours before surgery
  In the preoperative period, the patient's additional diseases, medications used, surgical history, and ASA score will be recorded.
Postoperative data | 24 hours after surgery
  The patient's general condition before discharge, and any complications related to surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Miray G Özdemir, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No